CLINICAL TRIAL: NCT01699932
Title: A Multinational, Open Label, Non Comparative, 24-week Study to Evaluate the Blood Glucose Lowering Efficacy and Safety of a Fixed Dose Combination of Glimepiride and Metformin in Patients With Inadequately Controlled Type 2 Diabetes
Brief Title: Efficacy and Safety of the Fixed Dose Combination of Glimepiride+Metformin in Type 2 Diabetic Patients Inadequately Controlled
Acronym: LEGEND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLMET_R_05823; U1111-1120-0058 (Other: UTN)
Record Dates: First submitted 2012-09-26; First posted 2012-10-04 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): 24-week treatment period: starting dose will be of 2/1000 mg or 4/2000 mg of glimepiride/metformin fixed combination (Amaryl M® ) depending on the previous treatment and dose. The Interventional medicinal product's dose will be increased every 2 weeks up to the maximum tolerated dose of 8/2000 mg of Amaryl M® , and adjusted throughout the 24-week treatment period according to fasting Self Monitored Plasma Glucose (SMPG) values in the objective to obtain fasting SMPG values ≤ 130mg/dL (7.2mmol/L) and > 70 mg/dL (3.9mmol/L) without symptomatic hypoglycemia.
  Interventions: Drug: Glimepiride+metformin (Amaryl M®) - HOE4900

INTERVENTIONS:
Drug: Glimepiride+metformin (Amaryl M®) - HOE4900 — Pharmaceutical form:tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

-To demonstrate the efficacy of a fixed combination of glimepiride + metformin in terms of HbA1c reduction, during 24-week treatment period in patients with inadequately controlled type 2 diabetes mellitus.

Secondary Objective:

To assess the effects of the fixed combination of glimepiride and metformin at week 24 on:

* Percentage of patients reaching HbA1c <7%
* Percentage of patients reaching HbA1c <6.5%.
* Fasting Plasma Glucose (FPG)
* Safety and tolerability

DETAILED DESCRIPTION:
The study duration for each patient is approximately 27 weeks with 3 periods: 2-week screening period followed by 24-week treatment period and 3 days follow-up period with a last call phone visit.

ELIGIBILITY:
Inclusion criteria:

* Patients with type 2 diabetes mellitus inadequately controlled despite a treatment with sulfonylurea (SU) alone or metformin alone or a free combination of SU and metformin prior to the study entry.
* Signed informed consent, obtained prior any study procedure

Exclusion criteria:

* Age < legal age of adulthood
* HbA1c < 7% or ≥ 11%
* BMI > 35 kg/m2
* Treatment with a stable dose of maximally tolerated SU alone or metformin alone or the free combination of SU and metformin for less than 12 weeks prior to the screening visit.
* Patients who received any anti-diabetic drug other than SU or metformin within 12 weeks prior to the screening visit.
* Diabetes other than type 2 diabetes (e.g. type 1 diabetes, diabetes secondary to pancreatic disorders, drug or chemical agent intake…)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | from baseline to week 24

SECONDARY OUTCOMES:
Percentage of patients with HbA1c < 7% | at week 24
Percentage of patients with HbA1c < 6.5% | at week 24
Change in Fasting Plasma Glucose (FPG) | from baseline to week 24
Number of patients with adverse events | over the 24-week treatment period
Hypoglycemia | over the 24-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- Lebanon (2):
  - Investigational Site Number 422-002, Beirut
  - Investigational Site Number 422-001, Hazmiyeh
- Russia (3):
  - Investigational Site Number 643-03, Saint Petersburg
  - Investigational Site Number 643002, Saint Petersburg
  - Investigational Site Number 643001, Samara
- Ukraine (8):
  - Investigational Site Number 804003, Chernivtsi
  - Investigational Site Number 804008, Donetsk
  - Investigational Site Number 804004, Donetsk
  - Investigational Site Number 804001, Donetsk
  - Investigational Site Number 804010, Odesa
  - Investigational Site Number 804006, Poltava
  - Investigational Site Number 804007, Vinnytsia
  - Investigational Site Number 804002, Vinnytsia